CLINICAL TRIAL: NCT01766648
Title: A Multicentre, Randomized Trial of Far Cortical Locking Versus Standard Constructs for Acute, Displaced Fractures of the Distal Femur Treated With Locked Plate Fixation
Brief Title: Far Cortical Locking Versus Standard Constructs for Distal Femur Fractures
Acronym: FCL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kelly A. Lefaivre, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H12-03489
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Distal Femur Fracture
Keywords: Distal; Femur; Locking; Screw; Fracture; Healing
MeSH Terms: conditions — Femoral Fractures, Distal; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Far Cortical Locking screw fixation (Experimental): Far Cortical Locking screw fixation
  Interventions: Device: Far Cortical locking screw fixation
- Standard screw fixation (Active Comparator): Standard screw fixation
  Interventions: Device: Standard screw fixation

INTERVENTIONS:
Device: Far Cortical locking screw fixation — Standard screw fixation
  Arms: Far Cortical Locking screw fixation
Device: Standard screw fixation
  Arms: Standard screw fixation

SUMMARY:
To determine if Far Cortical Locking screws increase fracture healing rates at 3 months in Closed Distal Femur Fractures in adults when compared to Standard screw constructs.

Fracture healing at 3 months will be assessed via radiographic and clinical assessment of the fracture.

Null Hypothesis: There will be no difference in fracture healing at 3 months post-fixation between subjects treated with far cortical locking screw or standard screw fixation.

DETAILED DESCRIPTION:
A multicentre randomized controlled trial with a sample size of 138 subjects.

Primary Outcome is fracture healing at 3 months via radiographic and and clinical assessment.

Radiographic healing will be defined as bridging of one or more cortices as seen on x-ray. Radiographic assessment will be centrally adjudicated by a committee of three study investigators.

Clinical healing will be assessed using the Function Index for Trauma (FIX-IT).

Secondary outcome measurements will include patient-reported quality of life and CT quantification of fracture callus volume.

Quality of life will be measured with the Short-Form 36 Version 2 (SF-36) instrument at all follow-up intervals.

A CT scan of the fracture site will be performed at the 3 month follow-up. Using a quantitative protocol the volume of callus will be measured and the extent of cortical bridging will be assessed.

Additional secondary outcomes include radiographic and clinical healing, as well as patient-important complications. These will include adverse events, delayed union (>6 months), non union (failure for fracture healing to progress on serial x-rays between 6 and 9 months), malalignment (>5 degrees), hardware failure, infection, and reoperation. Information surrounding the type of complication, duration, management and/or treatment of all complications will be recorded

A Data Safety Monitoring Board will be established to independently monitor trial data.

Specific inclusion criteria:

* Men or women ages 18 years or older
* Displaced distal femur fracture (OTA 33A or 33C) as seen in radiographs
* Planned treatment using a distal femur locking plate
* Ability to read and speak English or availability of translator willing to assist with completion of study forms
* Fractures < 14 days post injury
* Provision of informed consent

Specific exclusion criteria:

* Open distal femur fracture requiring flap or vascular repair (grade 3b or 3c)
* Planned fixation strategy includes interfragmentary lag fixation of non-articular fractures
* Active local infection
* Limited life expectancy due to significant medical co-morbidity or medical contraindication to surgery
* Inability to comply with rehabilitation or form completion
* Likely problems, in the judgment of the investigators, with maintaining follow-up (i.e. patients with no fixed address, patients not mentally competent to give consent, etc.)
* Non-ambulatory patients
* Lack of bone substance or poor bone quality which, in the surgeon's judgment, makes locked plate fixation impossible
* Periprosthetic fractures
* Any concomitant lower-extremity injury that requires non-weight-bearing beyond 6 weeks post-operative
* Addition of bone graft, bone graft substitute or BMP
* Pregnant women

ELIGIBILITY:
Specific inclusion criteria:

* Men or women ages 18 years or older
* Displaced distal femur fracture (OTA 33A or 33C) as seen in radiographs
* Planned treatment using a distal femur locking plate
* Ability to read and speak English or availability of translator willing to assist with completion of study forms
* Fractures < 14 days post injury
* Provision of informed consent

Specific exclusion criteria:

* Open distal femur fracture requiring flap or vascular repair (grade 3b or 3c)
* Planned fixation strategy includes interfragmentary lag fixation of non-articular fractures
* Active local infection
* Limited life expectancy due to significant medical co-morbidity or medical contraindication to surgery
* Inability to comply with rehabilitation or form completion
* Likely problems, in the judgment of the investigators, with maintaining follow-up (i.e. patients with no fixed address, patients not mentally competent to give consent, etc.)
* Non-ambulatory patients
* Lack of bone substance or poor bone quality which, in the surgeon's judgment, makes locked plate fixation impossible
* Periprosthetic fractures
* Any concomitant lower-extremity injury that requires non-weight-bearing beyond 6 weeks post-operative
* Addition of bone graft, bone graft substitute or BMP
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Composite fracture healing | 3 months
  Radiographic fracture healing defined as bridging of 1 or more cortices. Clinical fracture healing assessed with FIX-IT.
  Using the win ratio method, we hierarchically assessed radiographic healing, followed by clinical fracture healing. The pairwise comparison proceeds in a hierarchical fashion, using radiographic healing, followed by the FIX-IT score when patients cannot be differentiated based on radiographic healing. For each pairwise comparison, the treatment groups are assigned a win, loss, or tie. We calculate the win ratio as the number of wins in the FCL screw treatment group divided by the number of wins in the Standard screw group.

SECONDARY OUTCOMES:
Radiographic healing | 3 months
  Union is defined as the bridging of 1 or more cortices with stable fixation by three months post-fixation.
Clinical healing | 3 months
  We assessed clinical fracture healing using the Function Index for Trauma (FIX-IT) score. The FIX-IT instrument quantifies clinical healing by aggregating a 0- to 6-point assessment of weight-bearing and fracture site pain for a maximum score of 12 points, indicating the highest level of functional healing.
Patient-reported health-related quality of life | 3 months
  Assessment of SF-36 scores (physical component and mental component)
Patient-reported health-related quality of life | 12 months
  Assessment of SF-36 scores (physical component and mental component)
CT quantification of fracture callus volume | 3 months
  Using a quantitative protocol, the volume of callus will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Lefaivre, MD, Principal Investigator — University of British Columbia, Vancouver Coastal Health Authority
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Claireaux HA, Searle HKC, Parsons NR, Griffin XL. Interventions for treating fractures of the distal femur in adults. Cochrane Database Syst Rev. 2022 Oct 5;10(10):CD010606. doi: 10.1002/14651858.CD010606.pub3. PMID 36197809